CLINICAL TRIAL: NCT01346514
Title: Addiction Housing Case Management for Homeless Veterans Enrolled in Addictions Treatment
Brief Title: Addiction Housing Case Management for Homeless Veterans
Acronym: AHCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SDR 11-231
Record Dates: First submitted 2011-04-29; First posted 2011-05-03 (Estimated); Results first posted 2017-02-28 (Actual); Last update posted 2017-02-28 (Actual); Status verified 2017-01

CONDITIONS: Homelessness; Substance Abuse Disorders; Mental Disorders
Keywords: Homeless Persons; Housing; Case Management; Veterans; Substance Related Disorders; Mental Disorders; Social Adjustment
MeSH Terms: conditions — Mental Disorders; Substance-Related Disorders; Social Adjustment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Addiction/Housing Case Management(AHCM) (Experimental): The AHCM condition provided individual case management, delivered at the VA and in the community, designed to assist homeless Veterans with SUD issues who may be unable to take advantage of housing opportunities available in the VA due to difficulty navigating multiple services and maintaining stability with respect to SUD and co-occurring mental health conditions.
  Interventions: Behavioral: Intensive Addiction/Housing Case Management
- Arm 2: Housing Support Group(HSG) (Active Comparator): The HSG condition involved a weekly drop-in housing support group.
  Interventions: Behavioral: Housing Support Group

INTERVENTIONS:
Behavioral: Intensive Addiction/Housing Case Management — AHCM provided: 1) support in obtaining/maintaining housing through education about resources, coordination with VA and community housing program providers, assistance in establishing housing program eligibility, and problem-solving around threats to housing stability; 2) support for SUD and related issues that affect housing status through treatment engagement/re-engagement, referrals for needed services (e.g. psychiatric, medical, vocational), and addressing substance use issues proactively; 3) promotion of residential stability through Life Skills Training, which was designed to improve key skills (room and self-care, money management, and community participation).
  Other Names: AHCM
  Arms: Arm 1: Addiction/Housing Case Management(AHCM)
Behavioral: Housing Support Group — The HSG focused on gaining support from fellow study participants and learning from those who successfully obtained housing. Group facilitators provided education about housing resources and assistance with housing-related issues.
  Other Names: HSG
  Arms: Arm 2: Housing Support Group(HSG)

SUMMARY:
The study examined intensive case management for homeless Veterans in addiction treatment by integrating addiction/housing case managers (AHCM), operating from a Life Skills Training perspective, into an addiction specialty program. The primary aim was to determine whether the AHCM intervention increases number of days housed during the year following treatment entry. Secondary aims were to compare costs and cost-effectiveness of AHCM vs. time and attention control, determine if AHCM improves addiction outcomes and functional status, and examine treatment process variables associated with improved outcomes.

DETAILED DESCRIPTION:
Background: Homelessness, substance use, and co-occurring psychiatric disorders form a mutually perpetuating, downwardly spiraling triad that maintains a state of homelessness, increases morbidity and mortality and thereby escalates health care utilization and costs. Addiction treatment is one portal of health care entry accessed by many Veterans with this devastating triad, yet addiction treatment fails to address homelessness directly. Homeless Veterans entering addiction treatment have worse treatment outcomes and incur more costs than housed Veterans entering such treatment. Further, many homeless Veterans never obtain housing after treatment entry and substantial proportion of those who do may subsequently return to homelessness. Assertive community treatment / intensive case management shows promise in improving housing status, as well as substance use and mental health outcomes in this population. Life Skills Training, which has been shown to improve the likelihood of maintaining housing, may increase the effectiveness of this method of treatment. An approach to homelessness incorporating assertive community treatment / intensive case management and Life Skills Training has never previously been integrated into VA addiction specialty care.

Objectives: The proposed study will examine intensive case management for homeless Veterans in addiction treatment by integrating addiction/housing case managers (AHCM), operating from a Life Skills Training perspective, into an addiction specialty program. The primary aim is to determine whether the AHCM intervention increases number of days housed during the year following treatment entry. Secondary aims are to compare costs and cost-effectiveness of AHCM vs. time and attention control, determine if AHCM improves addiction outcomes and functional status, and examine treatment process variables associated with improved outcomes.

Methods: The proposed study is a, parallel design, intention to treat, randomized clinical trial comparing the AHCM intervention to a time and attention control (weekly housing group) among homeless Veterans (N=400) newly entering addiction treatment. Following baseline assessment, Veterans will be randomly assigned, stratified by gender and primary substance problem, to one of the two treatment conditions and followed for 12 months. All Veterans will receive addiction treatment as usual. Veterans assigned to the AHCM condition will have a case manager who is integrated with the interdisciplinary treatment team. The AHCM will meet with the Veteran weekly, assist the Veteran with potential housing options, support the Veteran in continuing addiction treatment and psychiatric care, visit the Veteran in the community when appropriate, and obtain point of care urine toxicology testing to assess abstinence with the goal of addressing substance use issues proactively. The AHCM will educate the Veteran on needed basic life skills using existing manuals. Veterans assigned to the control condition will attend a weekly housing group where housing options are discussed. Participants will complete research assessments every 3 months through one year and then every 6 months for up to 2 years post-randomization to assess housing status and other outcomes. The Northwest Regional Data Warehouse and Decision Support System data sources will be used to determine outpatient and inpatient VA health care services and costs for the 1 year before and 2 years after study enrollment.

Impact: If the AHCM model interrupts the mutually perpetuating triad of homelessness, substance use, and co-occurring psychiatric disorders by increasing days stably housed, reducing costs and excessive health care utilization, and improving functional status, the model could be feasibly and rapidly replicated in VA addiction programs nationwide thereby decreasing homelessness among Veterans and preserving precious health care resources.

ELIGIBILITY:
Inclusion Criteria:

* Veterans newly presenting or returning to specialty treatment for substance dependence at VA Puget Sound Seattle Division who, after an initial evaluation, are scheduled for a treatment appointment in the Addiction Treatment Center
* Currently homeless (unsheltered, staying in temporary emergency shelter, or doubled up with friends/family)

Exclusion Criteria:

* Not planning to stay in the Puget Sound area during the next 12 months
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2011-10; Primary Completion 2015-11 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J. Saxon, MD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Malte CA, Cox K, Saxon AJ. Providing intensive addiction/housing case management to homeless veterans enrolled in addictions treatment: A randomized controlled trial. Psychol Addict Behav. 2017 May;31(3):231-241. doi: 10.1037/adb0000273. PMID 28481614
- [Derived] Cox KB, Malte CA, Saxon AJ. Characteristics and service utilization of homeless veterans entering VA substance use treatment. Psychol Serv. 2017 May;14(2):208-213. doi: 10.1037/ser0000133. PMID 28481606

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (n=181) were recruited from the VA Puget Sound, Seattle Division between October 2011 and November 2015.
Groups:
- Arm 1/Addiction Housing Case Management (AHCM): AHCM intervention/ AHCM involves intensive case management for housing, substance use, and related issues. Veterans assigned to the AHCM condition will have a case manager who is integrated with the interdisciplinary treatment team. The AHCM will meet with the Veteran weekly, assist the Veteran with potential housing options, support the Veteran in continuing addiction treatment and psychiatric care, visit the Veteran in the community when appropriate, and obtain point of care urine toxicology testing to assess abstinence with the goal of addressing substance use issues proactively. The AHCM will educate the Veteran on needed basic life skills using existing manuals
- Arm 2/Housing Support Group (HSG): HSG/ The Housing Support Group is a time and attention control. Veterans assigned to HSG attend a weekly drop-in housing group where housing options are discussed and participants receive support from one another.
Period: Overall Study
Arm/Group | Arm 1/Addiction Housing Case Management (AHCM) | Arm 2/Housing Support Group (HSG)
Started | 91 | 90
3 Month Assessment | 83 | 68
6 Month Assessment | 74 | 61
9 Month Assessment | 67 | 59
12 Month Assessment | 62 | 53
Completed | 62 (Number of patients completing BL-12 months) | 53 (Number of patients completing BL-12 months.)
Not Completed | 29 | 37
Not completed — Lost to Follow-up | 19 | 30
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Death | 3 | 4

BASELINE CHARACTERISTICS:
Population: Participants were eligible to participate if they 1) were homeless (i.e. on the streets, in emergency shelter or doubled up without paying rent) ; 2) initiated a new substance use treatment episode within 30 days; and 3) intended to reside locally for one year.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1/Addiction Housing Case Management (AHCM) | Arm 2/Housing Support Group (HSG) | Total
Number analyzed (Participants) | 91 | 90 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (9.5) | 50.9 (9.6) | 50.9 (9.5)
Gender [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 89 | 88 | 177
Race/Ethnicity, Customized [Number; unit: participants]
  White | 55 | 53 | 108
  Black | 32 | 28 | 60
  Native American | 0 | 6 | 6
  Asian/Pacific Islander | 2 | 0 | 2
  Hispanic | 2 | 3 | 5
Primary Substance of Use [Number; unit: participants]
  Alcohol | 57 | 59 | 116
  Cocaine | 15 | 15 | 30
  Opioids | 9 | 8 | 17
  Other | 10 | 8 | 18
Time Homeless, Current Episode [Number; unit: participants]
  Less than 1 month | 15 | 10 | 25
  1-6 months | 31 | 27 | 58
  6-12 months | 21 | 15 | 36
  1-2 years | 9 | 10 | 19
  2 or more years | 15 | 27 | 42
  Unknown | 0 | 1 | 1
Episodes of Homelessness [Number; unit: participants]
  1 episode | 51 | 55 | 106
  2 episodes | 24 | 17 | 41
  3 episodes | 4 | 10 | 14
  4 episodes | 4 | 4 | 8
  5 or more episodes | 8 | 3 | 11
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Days Housed in AHCM vs. HSG, Baseline to 12 Months.
Description: The primary aim is to determine whether the Addiction/Housing Case Management intervention increases percent days in long-term housing (permanent or long-term transitional) during the year following treatment entry relative to a Housing Support Group.
Time Frame: 12 months (18 to 24 month outcomes examined in secondary analyses)
Population: The percent of days in long-term transitional housing and/or own home was calculated for all patients using self-report and VA Homeless Operations Management and Evaluation System (HOMES) data. Individuals with no self-report or HOMES data were coded as not housed.
Measure: Mean (95% Confidence Interval); unit: percent days housed
Groups:
- Arm 1/Addiction Housing Case Management (AHCM): The AHCM condition provided individual case management, delivered at the VA and in the community, designed to assist homeless Veterans with SUD issues. Case management focused on : 1) support in obtaining/maintaining housing through education about resources, coordination with VA and community housing program providers, assistance in establishing housing program eligibility, and problem-solving around threats to housing stability; 2) support for SUD and related issues that affect housing status through treatment engagement/re-engagement, referrals for needed services (e.g. psychiatric, medical, vocational), and addressing substance use issues proactively; 3) promotion of residential stability through Life Skills Training, which was designed to improve key skills (room and self-care, money management, and community participation).
- Arm 2/Housing Support Group (HSG): The HSG condition involved a weekly drop-in housing support group. The HSG focused on gaining support from fellow study participants and learning from those who successfully obtained housing. Group facilitators provided education about housing resources and assistance with housing-related issues.
Arm/Group | Arm 1/Addiction Housing Case Management (AHCM) | Arm 2/Housing Support Group (HSG)
Number analyzed (Participants) | 91 | 90
percent days housed
  Percent Days Housed, Baseline | 14.7 [9.3 to 20.2] | 12.0 [7.0 to 16.9]
  Percent Days Housed, 3 Month | 25.0 [18.1 to 31.8] | 14.1 [8.9 to 19.4]
  Percent Days Housed, 6 Month | 48.9 [39.6 to 58.2] | 44.4 [35.4 to 53.4]
  Percent Days Housed, 9 Month | 53.9 [44.3 to 63.5] | 48.5 [38.9 to 58.2]
  Percent Days Housed, 12 Month | 53.1 [43.3 to 62.8] | 51.4 [41.4 to 61.4]

2. Secondary Outcome: Costs and Cost-effectiveness of AHCM vs. HSG, Baseline to 12 Months
Description: Costs and cost-effectiveness of Addiction/Housing Case Management to the Housing Support Group condition.
Time Frame: Baseline to 12 months
Population: These analyses were not completed due to the lack of differences seen in the primary study outcomes (percent days housed) and quality of life measures (SF-36).
Groups:
- Arm 1: Addiction/Housing Case Management(AHCM): The AHCM condition provided individual case management, delivered at the VA and in the community, designed to assist homeless Veterans with SUD issues. Case management focused on : 1) support in obtaining/maintaining housing through education about resources, coordination with VA and community housing program providers, assistance in establishing housing program eligibility, and problem-solving around threats to housing stability; 2) support for SUD and related issues that affect housing status through treatment engagement/re-engagement, referrals for needed services (e.g. psychiatric, medical, vocational), and addressing substance use issues proactively; 3) promotion of residential stability through Life Skills Training, which was designed to improve key skills (room and self-care, money management, and community participation).
- Arm 2: Housing Support Group(HSG): The HSG condition involved a weekly drop-in housing support group. The HSG focused on gaining support from fellow study participants and learning from those who successfully obtained housing. Group facilitators provided education about housing resources and assistance with housing-related issues.
Arm/Group | Arm 1: Addiction/Housing Case Management(AHCM) | Arm 2: Housing Support Group(HSG)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Functional Status in AHCM vs. HSG From Baseline to 12 Months
Description: Determine if Addiction/Housing Case Management compared to a Housing Support Group control significantly improved functional status outcomes among homeless Veterans entering addiction specialty care over the 12-month study course. Functional status was measured by Medical, Employment, Family/Social, and Legal Composite Scores (range 0 to 1 with higher scores indicating greater severity) on the Addiction Severity Index (ASI) and the Physical Component Summary (PCS, range 0 to 100 with lower scores indicating greater severity) on the SF-36. Negative change on the ASI measures indicates improvement. Positive change on the SF-36 PCS indicates improvement.
Time Frame: Baseline to 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1/Addiction Housing Case Management (AHCM) | Arm 2/Housing Support Group (HSG)
Number analyzed (Participants) | 91 | 90
units on a scale
  ASI Medical Composite, Change BL to Month 12 | -0.05 [-0.16 to 0.05] | 0.04 [-0.06 to 0.14]
  ASI Employment Composite, Change BL to Month 12 | -0.05 [-0.10 to 0.00] | 0.00 [-0.05 to 0.04]
  ASI Family Composite, Change BL to Month 12 | -0.04 [-0.07 to 0.00] | -0.04 [-0.07 to -0.01]
  ASI Legal Composite, Change BL to Month 12 | -0.07 [-0.11 to -0.03] | -0.07 [-0.10 to -0.03]
  SF-36 Physical Component Summ, Chg BL to Month 12 | 0.89 [-1.09 to 2.87] | -1.07 [-3.04 to 0.91]

4. Secondary Outcome: Change in Alcohol and Drug Outcomes in AHCM vs. HSG From Baseline to 12 Months
Description: Determine if Addiction/Housing Case Management compared to a Housing Support Group control significantly improved alcohol and drug outcomes, as measured by Alcohol and Drug Composite Scores (range 0 to 1, with higher scores indicating greater severity) on the Addiction Severity Index (ASI), among homeless Veterans entering addiction specialty care over the 12-month study course. Negative change on the ASI measures indicates improvement.
Time Frame: Baseline to 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1: Addiction/Housing Case Management(AHCM) | Arm 2: Housing Support Group(HSG)
Number analyzed (Participants) | 91 | 90
units on a scale
  ASI Alcohol Composite, Change BL to Month 12 | -0.06 [-0.13 to 0.01] | -0.20 [-0.26 to -0.13]
  ASI Drug Composite, Change BL to Month 12 | -0.04 [-0.07 to -0.02] | -0.05 [-0.07 to -0.03]

5. Secondary Outcome: Change in Percent of Participants Abstinent From Baseline to 12 Month Follow-up
Description: Determine if Addiction/Housing Case Management compared to a Housing Support Group control significantly increase the percent of participants abstinent from alcohol and drugs over the past 30 days among homeless Veterans entering addiction specialty care over the 12-month study course. Positive change indicates improvement.
Time Frame: Baseline to 12 months
Measure: Number (95% Confidence Interval); unit: precentage of participants
Arm/Group | Arm 1/Addiction Housing Case Management (AHCM) | Arm 2/Housing Support Group (HSG)
Number analyzed (Participants) | 91 | 90
precentage of participants | 27.0 [12.2 to 41.7] | 30.5 [16.2 to 44.8]

6. Secondary Outcome: Change in Mental Health Status in AHCM vs. HSG From Baseline to 12 Months
Description: Determine if Addiction/Housing Case Management compared to a Housing Support Group control significantly improved mental health outcomes, as measured by the Psychiatric Composite Score (range 0 to 1, with higher scores indicating greater severity) on the Addiction Severity Index (ASI) and the Mental Component Summary (MCS, range 0 to 100 with lower scores indicating greater severity) of the SF-36, among homeless Veterans entering addiction specialty care over the 12-month study course. Negative change on the ASI Psychiatric Composite Score indicates improvement. Positive change on the SF-36 MCS indicates improvement.
Time Frame: Baseline to 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Arm 1: Addiction/Housing Case Management(AHCM) | Arm 2: Housing Support Group(HSG)
Number analyzed (Participants) | 91 | 90
units on a scale
  ASI Psychiatric Composite, Change BL to Month 12 | -0.11 [-0.17 to -0.04] | -0.13 [-0.19 to -0.07]
  SF-36 MCS, Change BL to Month 12 | 1.08 [-1.92 to 4.08] | 3.09 [0.63 to 5.55]

7. Secondary Outcome: Treatment Process Measures (Number of Treatment Sessions, Type of Housing Placement, and Change in Life Skills)
Description: Analyses will explore whether treatment process variables mediate differences in outcomes between Addiction/Housing Case Management and time and attention conditions.
Time Frame: Baseline to 12 months
Population: Due to the lack of differences seen in the primary housing outcomes between the AHCM and HSG conditions, tests of mediation were not completed.
Arm/Group | Arm 1: Addiction/Housing Case Management(AHCM) | Arm 2: Housing Support Group(HSG)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to 12 months.
Description: Data on hospitalizations and suicide attempts were collected from participant self-report and from VA medical record review at every assessment. Information on death was collected from medical record review and from the Vital Status file. Information on cause of death was not available. Information on non-serious adverse events were not collected.
Arm/Group | Arm 1/Addiction Housing Case Management (AHCM) | Arm 2/Housing Support Group (HSG)
Serious Adverse Events (participants affected / at risk) | 39/91 | 31/90
Other Adverse Events (participants affected / at risk) | 18/91 | 13/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1/Addiction Housing Case Management (AHCM) (N=91) | Arm 2/Housing Support Group (HSG) (N=90)
Death (General disorders) | 3 (3) | 4 (4)
Medical Hospitalization (General disorders) | 19 (36) | 16 (27) — Number of patients hospitalized on an acute medical unit between baseline and month 12.
Suicide attempt (Psychiatric disorders) | 2 (2) | 3 (6) — Number of patients with suicide attempt between baseline and month 12
Psychiatric Hospitalization (Psychiatric disorders) | 20 (35) | 8 (21) — Number of patients hospitalized on an acute psychiatric unit between baseline and month 12.
Inpatient Detoxification (Psychiatric disorders) | 11 (17) | 12 (22) — Number of patients hospitalized for alcohol/drug detoxification between baseline and month 12.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1/Addiction Housing Case Management (AHCM) (N=91) | Arm 2/Housing Support Group (HSG) (N=90)
Incarceration (Social circumstances) | 18 (34) | 13 (17) — Number of patients incarcerated between baseline and month 12

LIMITATIONS AND CAVEATS:
Study limitations include lower than expected recruitment, conducted at a single VA facility, research staff members were not blinded to study condition after baseline, high attrition rates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No